CLINICAL TRIAL: NCT00329420
Title: A Multi-center, Open-label Study to Investigate the Efficacy and Safety of CDP870 in Active Crohn's Disease Patients, Who Showed no Clinical Efficacy in a Remission Induction Study (Study C87037) But Showed Clinical Efficacy After Additional Remission Induction Therapy Was Applied, at Week 26 After Subcutaneous Administration of CDP870 400 mg From Week 8 Until Week 24 at 4-week Intervals
Brief Title: Maintenance Study Including Re-induction Therapy for Patients Who Did Not Show a Clinical Effect in Study C87037 (NCT00291668)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87048; 2014-004400-30 (EudraCT Number)
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Results first posted 2009-11-10 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; CDP870; Certolizumab pegol; CZP
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CZP 400 mg / Placebo (Experimental): Certolizumab pegol (CZP) 400 mg in this extension study / Placebo in double-blind main study (NCT00291668)
  Interventions: Biological: Certolizumab pegol
- CZP 400 mg / CZP 200 mg (Experimental): Certolizumab pegol (CZP) 400 mg in this extension study / Certolizumab pegol (CZP) 200 mg in double-blind main study (NCT00291668)
  Interventions: Biological: Certolizumab pegol
- CZP 400 mg / CZP 400 mg (Experimental): Certolizumab pegol (CZP) 400 mg in this extension study / Certolizumab pegol (CZP) 400 mg in double-blind main study (NCT00291668)
  Interventions: Biological: Certolizumab pegol

INTERVENTIONS:
Biological: Certolizumab pegol — Certolizumab pegol (CZP) 400 mg administered subcutaneously in a liquid formulation at Weeks 8, 10, 12, 16, 20, 24, 28 and 32 relative to the start of the 6-week double-blind main study C87037 (NCT00291668) where subjects received Placebo at Weeks 0, 2 and 4.
  Other Names: CDP870; Cimzia; CZP
  Arms: CZP 400 mg / Placebo
Biological: Certolizumab pegol — Certolizumab pegol (CZP) 400 mg administered subcutaneously in a liquid formulation at Weeks 8, 10, 12, 16, 20, 24, 28 and 32 relative to the start of the 6-week double-blind main study C87037 (NCT00291668) where subjects received Certolizumab pegol (CZP) 200 mg at Weeks 0, 2 and 4.
  Other Names: CDP870; Cimzia; CZP
  Arms: CZP 400 mg / CZP 200 mg
Biological: Certolizumab pegol — Certolizumab pegol (CZP) 400 mg administered subcutaneously in a liquid formulation at Weeks 8, 10, 12, 16, 20, 24, 28 and 32 relative to the start of the 6-week double-blind main study C87037 (NCT00291668) where subjects received Certolizumab pegol (CZP) 400 mg at Weeks 0, 2 and 4.
  Other Names: CDP870; Cimzia; CZP
  Arms: CZP 400 mg / CZP 400 mg

SUMMARY:
This 26-week extension study evaluates the efficacy and safety of certolizumab pegol administered subcutaneously every 4 weeks (dosed at Weeks 16, 20, 24, 28 and 32) in subjects with active Crohn's disease who had no clinical response at Week 6 to induction therapy in the 6-week double-blind main study, C87037 (NCT00291668), but subsequently showed clinical response at Week 14 to repeated induction therapy (dosed at Weeks 8, 10 and 12) in this extension study.

DETAILED DESCRIPTION:
This study is an open-label extension study which follows on from the 6-week double-blind main study C87037 (NCT00291668). All 'Week' numbers quoted are relative to the start of the double-blind main study. The first visit in this extension study is at Week 8, and the final efficacy assessment in this extension study, 26 weeks later, is at Week 34.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who gave written informed consent and who did not show clinical efficacy at Week 6 of the double-blind main study (NCT00291668) [reduction in Crohn's Disease Activity Index (CDAI) score of ≥100 points from Week 0, or remission (CDAI ≤150)]

Exclusion Criteria:

* Subjects who experienced aggravation of Crohn's Disease during the double-blind main study (NCT00291668) and required treatment change

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2006-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (23):
- Japan (23):
  - Aichi-Gun, Aichi-ken
  - Nagoya, Aichi-ken
  - Toyoake, Aichi-ken
  - Toyohashi, Aichi-ken
  - Kashiwa, Chiba
  - Sakura, Chiba
  - Chikusino, Fukuoka
  - Fukuoka, Fukuoka
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Kagoshima, Kagoshima-ken
  - Yokohama, Kanagawa
  - Miyazaki-gun, Miyazaki
  - Nagasaki, Nagasaki
  - Niigata, Niigata
  - Kurashiki, Okayama-ken
  - Tyuto-gun, Okianawa
  - Osaka, Osaka
  - Osaka Suita, Osaka
  - Shiga Otsu, Shiga
  - Shinjyuku/Tokyo, Tokyo
  - Shinjyuku, Tokyo

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-responders at Week 6 of the double-blind main study, C87037 (NCT00291668) could enter this single-group open-label extension study, C87048 (NCT00329420). Recruitment into this extension study was between May 2006 and May 2008. Of the 26 hospitals in the main study (NCT00291668), 16 sites went on to enter subjects into this extension study.
Pre-assignment Details: Subjects who responded to re-induction (Week 14 visit) in this extension study could enter the 4-weekly dosing phase. Efficacy data are based on these 26 subjects. However, adverse event data are based on all 46 subjects who entered this extension study. Data are presented by the three possible treatment sequences received across both studies.
Groups:
- CZP 400 mg / Placebo: Certolizumab pegol (CZP) 400 mg (3 doses 2-weekly then 5 doses 4-weekly) in this extension study / Placebo (3 doses 2-weekly) in the 6-week double-blind main study (NCT00291668)
- CZP 400 mg / CZP 200 mg: Certolizumab pegol (CZP) 400 mg (3 doses 2-weekly then 5 doses 4-weekly) in this extension study / Certolizumab pegol (CZP) 200 mg (3 doses 2-weekly) in the 6-week double-blind main study (NCT00291668)
- CZP 400 mg / CZP 400 mg: Certolizumab pegol (CZP) 400 mg (3 doses 2-weekly then 5 doses 4-weekly) in this extension study / Certolizumab pegol (CZP) 400 mg (3 doses 2-weekly) in the 6-week double-blind main study (NCT00291668)
Period: Re-induction Phase
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Started | 18 | 13 | 15
Completed | 12 (Completed = Reached Week 14 (end of re-induction phase) and responded to re-induction at that time.) | 7 (Completed = Reached Week 14 (end of re-induction phase) and responded to re-induction at that time.) | 7 (Completed = Reached Week 14 (end of re-induction phase) and responded to re-induction at that time.)
Not Completed | 6 | 6 | 8
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 1
Not completed — Did not respond to re-induction | 6 | 5 | 7
Period: 4-weekly Dosing Phase (Responders Only)
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Started | 12 | 7 | 7
Completed | 8 | 5 | 6
Not Completed | 4 | 2 | 1
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Withdrawal of Consent | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg | Total
Number analyzed (Participants) | 18 | 13 | 15 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 17 | 13 | 15 | 45
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (7.5) | 37.5 (8.2) | 29.9 (5.9) | 32.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 14 | 9 | 12 | 35
Region of Enrollment [Number; unit: participants]
  Japan | 18 | 13 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 34
Description: Crohn's disease activity index (CDAI) responders are subjects achieving either clinical response (a reduction in CDAI score of ≥100 points from Week 0), or remission (CDAI ≤150). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
Time Frame: Week 0 and Week 34 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 34' is 26 weeks after the first visit in this extension study.
Population: Non-responders at Week 6 of main study C87037 (NCT00291668) could enter this extension study, C87048 (NCT00329420). This summary is based on the 26 subjects in the Full Analysis Set (FAS) Population who responded to re-induction at Week 14. Subject withdrawal or use of rescue therapy is counted as non-response from that time onwards in that study.
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 66.7 | 28.6 | 42.9
  Percentage of CDAI non-responders | 33.3 | 71.4 | 57.1

2. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 8
Description: Crohn's disease activity index (CDAI) is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 0 and Week 8 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 8' is the first visit in this extension study.
Population: Please see under the primary endpoint for explanation of entry into this extension study, C87048 (NCT00329420), and of 26 subjects being in the subgroup of "Responders to Re-induction", based on the Full Analysis Set. All those in this subgroup with data are included in this summary.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | -20.5 (81.6) | -53.1 (38.1) | -63.8 (26.4)

3. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 10
Description: as for outcome 2
Time Frame: Week 0 and Week 10 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 10' is 2 weeks after the first visit in this extension study.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | -96.1 (76.1) | -100.3 (35.4) | -90.0 (18.2)

4. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 12
Description: as for outcome 2
Time Frame: Week 0 and Week 12 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 12' is 4 weeks after the first visit in this extension study.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | -101.3 (56.6) | -100.5 (49.3) | -109.9 (36.7)

5. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 14
Description: as for outcome 2
Time Frame: Week 0 and Week 14 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 14' is 6 weeks after the first visit in this extension study.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | -124.3 (50.4) | -131.7 (41.3) | -147.0 (45.2)

6. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 16
Description: as for outcome 2
Time Frame: Week 0 and Week 16 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 16' is 8 weeks after the first visit in this extension study.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | -121.0 (57.7) | -70.4 (84.1) | -136.2 (32.2)

7. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 20
Description: as for outcome 2
Time Frame: Week 0 and Week 20 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 20' is 12 weeks after the first visit in this extension study.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | -105.3 (82.9) | -79.6 (60.9) | -130.9 (62.5)

8. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 24
Description: as for outcome 2
Time Frame: Week 0 and Week 24 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 24' is 16 weeks after the first visit in this extension study.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | -89.8 (79.8) | -70.6 (91.3) | -150.2 (48.0)

9. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 28
Description: as for outcome 2
Time Frame: Week 0 and Week 28 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 28' is 20 weeks after the first visit in this extension study.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | -118.2 (62.6) | -67.3 (77.1) | -154.8 (74.2)

10. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 32
Description: as for outcome 2
Time Frame: Week 0 and Week 32 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 32' is 24 weeks after the first visit in this extension study.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 6
score on a scale | -89.0 (88.3) | -77.3 (70.9) | -128.3 (75.3)

11. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 34
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 5
score on a scale | -134.9 (39.3) | -97.4 (33.1) | -132.7 (89.7)

12. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: as for outcome 2
Time Frame: Week 0 and Last Visit (Week 34 relative to the start of the 6-week double-blind main study (NCT00291668) for completers or the Withdrawal Visit for premature withdrawals). 'Week 34' is 26 weeks after the first visit in this extension study.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 6 | 5
score on a scale | -112.0 (75.6) | -61.0 (93.7) | -132.7 (89.7)

13. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 8
Description: as for outcome 1
Time Frame: as for outcome 2
Population: Please see under the primary endpoint for explanation of entry into this extension study, C87048 (NCT00329420), and of 26 subjects being in the subgroup of "Responders to Re-induction", based on the Full Analysis Set. This also details withdrawal or rescue therapy being counted as non-response in a study from that time onwards in that study.
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 8.3 | 14.3 | 14.3
  Percentage of CDAI non-responders | 91.7 | 85.7 | 85.7

14. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 10
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 13
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 41.7 | 71.4 | 42.9
  Percentage of CDAI non-responders | 58.3 | 28.6 | 57.1

15. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 12
Description: as for outcome 1
Time Frame: as for outcome 4
Population: as for outcome 13
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 50.0 | 71.4 | 57.1
  Percentage of CDAI non-responders | 50.0 | 28.6 | 42.9

16. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 14
Description: as for outcome 1
Time Frame: as for outcome 5
Population: as for outcome 13
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 100.0 | 100.0 | 100.0
  Percentage of CDAI non-responders | 0.0 | 0.0 | 0.0

17. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 16
Description: as for outcome 1
Time Frame: as for outcome 6
Population: as for outcome 13
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 66.7 | 42.9 | 85.7
  Percentage of CDAI non-responders | 33.3 | 57.1 | 14.3

18. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 20
Description: as for outcome 1
Time Frame: as for outcome 7
Population: as for outcome 13
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 41.7 | 28.6 | 85.7
  Percentage of CDAI non-responders | 58.3 | 71.4 | 14.3

19. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 24
Description: as for outcome 1
Time Frame: as for outcome 8
Population: as for outcome 13
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 41.7 | 57.1 | 71.4
  Percentage of CDAI non-responders | 58.3 | 42.9 | 28.6

20. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 28
Description: as for outcome 1
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 50.0 | 28.6 | 57.1
  Percentage of CDAI non-responders | 50.0 | 71.4 | 42.9

21. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 32
Description: as for outcome 1
Time Frame: as for outcome 10
Population: as for outcome 13
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 33.3 | 28.6 | 57.1
  Percentage of CDAI non-responders | 66.7 | 71.4 | 42.9

22. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: as for outcome 1
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of CDAI responders | 66.7 | 28.6 | 42.9
  Percentage of CDAI non-responders | 33.3 | 71.4 | 57.1

23. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 8
Description: Crohn's disease activity index (CDAI) is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
Time Frame: Week 8 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 8' is the first visit in this extension study.
Population: Please see under the primary endpoint for explanation of entry into this extension study, C87048 (NCT00329420), and of 26 subjects being in the subgroup of "Responders to Re-induction", based on the Full Analysis Set. If a subject withdrew or received rescue therapy, they were counted as not in remission in that study from that time-point onwards.
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 0.0 | 0.0 | 14.3
  Percentage of subjects not in remission | 100.0 | 100.0 | 85.7

24. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 10
Description: as for outcome 23
Time Frame: Week 10 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 10' is 2 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 33.3 | 42.9 | 14.3
  Percentage of subjects not in remission | 66.7 | 57.1 | 85.7

25. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 12
Description: as for outcome 23
Time Frame: Week 12 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 12' is 4 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 25.0 | 42.9 | 42.9
  Percentage of subjects not in remission | 75.0 | 57.1 | 57.1

26. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 14
Description: as for outcome 23
Time Frame: Week 14 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 14' is 6 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 66.7 | 71.4 | 71.4
  Percentage of subjects not in remission | 33.3 | 28.6 | 28.6

27. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 16
Description: as for outcome 23
Time Frame: Week 16 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 16' is 8 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 33.3 | 28.6 | 57.1
  Percentage of subjects not in remission | 66.7 | 71.4 | 42.9

28. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 20
Description: as for outcome 23
Time Frame: Week 20 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 20' is 12 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 33.3 | 28.6 | 57.1
  Percentage of subjects not in remission | 66.7 | 71.4 | 42.9

29. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 24
Description: as for outcome 23
Time Frame: Week 24 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 24' is 16 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 16.7 | 42.9 | 71.4
  Percentage of subjects not in remission | 83.3 | 57.1 | 28.6

30. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 28
Description: as for outcome 23
Time Frame: Week 28 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 28' is 20 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 25.0 | 28.6 | 57.1
  Percentage of subjects not in remission | 75.0 | 71.4 | 42.9

31. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 32
Description: as for outcome 23
Time Frame: Week 32 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 32' is 24 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 16.7 | 28.6 | 42.9
  Percentage of subjects not in remission | 83.3 | 71.4 | 57.1

32. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 34
Description: as for outcome 23
Time Frame: Week 34 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 34' is 26 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 33.3 | 28.6 | 42.9
  Percentage of subjects not in remission | 66.7 | 71.4 | 57.1

33. Secondary Outcome: Percentage of Subjects Achieving Remission at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: as for outcome 23
Time Frame: Last Visit (Week 34 relative to the start of the 6-week double-blind main study (NCT00291668) for completers or the Withdrawal Visit for premature withdrawals). 'Week 34' is 26 weeks after the first visit in this extension study.
Population: as for outcome 23
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
Percentage of subjects
  Percentage of subjects in remission | 33.3 | 28.6 | 42.9
  Percentage of subjects not in remission | 66.7 | 71.4 | 57.1

34. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the earliest of:
  * time to an increase from Week 14 of ≥100 points in Crohn's Disease Activity Index (CDAI) score and CDAI>175 points for at least 2 consecutive visits,
  * time to use of rescue therapy, or,
  * time to subject withdrawal from the study.
Time Frame: Week 14 to Week 34 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 14' is the visit at which response to re-induction is assessed and 'Week 34' is 26 weeks after the first visit in this extension study.
Population: Non-responders at Week 6 of Study C87037 (NCT00291668) could enter this extension study, C87048 (NCT00329420). As so few subjects experienced disease progression in this study it was not possible to calculate the median time to disease progression. Please see outcome measure 124 where the number of subjects with disease progression is presented.
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 8
Description: The IBDQ Global Score is the sum of 32 responses, each ranging from 0 to 7, thus the Global Score ranges from 0 to 224; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: Please see under the primary endpoint for explanation of entry into this extension study, C87048 (NCT00329420). Subjects who respond to re-induction in the Full Analysis Set with data at both time-points are included. Data collected after receipt of rescue therapy in a study have been set to missing in that study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 4.6 (15.3) | 9.1 (7.5) | 5.3 (13.8)

36. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 10
Description: as for outcome 35
Time Frame: as for outcome 3
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 17.0 (17.5) | 20.9 (24.9) | 15.1 (13.4)

37. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 12
Description: as for outcome 35
Time Frame: as for outcome 4
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 17.3 (12.0) | 26.3 (33.6) | 20.1 (16.6)

38. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 14
Description: as for outcome 35
Time Frame: as for outcome 5
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 20.1 (12.3) | 28.6 (22.9) | 26.3 (16.1)

39. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 16
Description: as for outcome 35
Time Frame: as for outcome 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 16.3 (12.2) | 15.3 (19.1) | 20.0 (16.4)

40. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 20
Description: as for outcome 35
Time Frame: as for outcome 7
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | 12.2 (16.0) | 18.4 (27.5) | 15.9 (14.7)

41. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 24
Description: as for outcome 35
Time Frame: as for outcome 8
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | 8.3 (14.5) | 7.6 (23.3) | 18.4 (18.0)

42. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 28
Description: as for outcome 35
Time Frame: as for outcome 9
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | 14.9 (20.0) | 11.4 (24.3) | 15.9 (19.3)

43. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 32
Description: as for outcome 35
Time Frame: as for outcome 10
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 6
score on a scale | 11.3 (17.8) | 11.2 (21.7) | 25.3 (17.0)

44. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 34
Description: as for outcome 35
Time Frame: as for outcome 1
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 5
score on a scale | 21.6 (16.9) | 14.8 (23.6) | 20.6 (17.6)

45. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score is the sum of 32 responses, each ranging from 0 to 7, thus the Global Score ranges from 0 to 224; a higher score indicating a better quality of life.
Time Frame: as for outcome 12
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 6 | 5
score on a scale | 15.6 (19.5) | 10.8 (23.3) | 20.6 (17.6)

46. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 8
Description: The IBDQ Bowel Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 1.9 (7.5) | 6.4 (5.6) | 2.4 (5.3)

47. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 10
Description: as for outcome 46
Time Frame: as for outcome 3
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 6.2 (8.4) | 10.6 (8.4) | 5.9 (7.1)

48. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 12
Description: as for outcome 46
Time Frame: as for outcome 4
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 5.7 (4.4) | 11.7 (9.7) | 7.4 (7.9)

49. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 14
Description: as for outcome 46
Time Frame: as for outcome 5
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 6.9 (5.6) | 12.3 (9.3) | 9.3 (7.0)

50. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 16
Description: as for outcome 46
Time Frame: as for outcome 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 5.2 (6.3) | 8.4 (9.9) | 6.3 (7.2)

51. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 20
Description: as for outcome 46
Time Frame: as for outcome 7
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | 3.5 (7.4) | 9.9 (11.7) | 5.1 (5.5)

52. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 24
Description: as for outcome 46
Time Frame: as for outcome 8
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | 0.7 (5.3) | 4.7 (11.0) | 5.6 (8.2)

53. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 28
Description: as for outcome 46
Time Frame: as for outcome 9
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | 4.6 (6.0) | 8.3 (10.0) | 5.4 (8.4)

54. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 32
Description: as for outcome 46
Time Frame: as for outcome 10
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 6
score on a scale | 3.1 (6.7) | 9.6 (11.0) | 7.5 (5.1)

55. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Week 34
Description: as for outcome 46
Time Frame: as for outcome 1
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 5
score on a scale | 7.1 (4.9) | 11.8 (9.8) | 5.8 (6.5)

56. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 12
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 6 | 5
score on a scale | 5.5 (6.9) | 8.3 (12.2) | 5.8 (6.5)

57. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 8
Description: The IBDQ Systemic Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 1.4 (3.4) | 0.6 (1.7) | 1.7 (1.6)

58. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 10
Description: as for outcome 57
Time Frame: as for outcome 3
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 4.6 (4.4) | 3.7 (6.2) | 3.9 (1.3)

59. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 12
Description: as for outcome 57
Time Frame: as for outcome 4
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 5.7 (3.2) | 5.0 (7.3) | 5.1 (2.1)

60. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 14
Description: as for outcome 57
Time Frame: as for outcome 5
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 5.9 (3.0) | 6.4 (4.3) | 6.3 (3.1)

61. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 16
Description: as for outcome 57
Time Frame: as for outcome 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 5.5 (2.4) | 3.9 (3.7) | 5.3 (3.5)

62. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 20
Description: as for outcome 57
Time Frame: as for outcome 7
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | 3.6 (4.0) | 3.6 (6.3) | 3.6 (2.6)

63. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 24
Description: as for outcome 57
Time Frame: as for outcome 8
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | 3.1 (2.9) | 2.1 (5.9) | 4.1 (2.7)

64. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 28
Description: as for outcome 57
Time Frame: as for outcome 9
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | 3.0 (6.1) | 3.0 (5.8) | 4.4 (3.6)

65. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 32
Description: as for outcome 57
Time Frame: as for outcome 10
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 6
score on a scale | 3.4 (4.3) | 0.4 (3.1) | 6.8 (3.8)

66. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Week 34
Description: as for outcome 57
Time Frame: as for outcome 1
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 5
score on a scale | 5.0 (3.2) | 3.0 (4.8) | 5.4 (2.1)

67. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 12
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 6 | 5
score on a scale | 4.2 (4.1) | 3.2 (4.4) | 5.4 (2.1)

68. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 8
Description: The IBDQ Emotional Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | -0.3 (6.1) | 2.1 (2.3) | 0.4 (6.7)

69. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 10
Description: as for outcome 68
Time Frame: as for outcome 3
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 3.3 (4.7) | 4.4 (9.7) | 4.3 (5.9)

70. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 12
Description: as for outcome 68
Time Frame: as for outcome 4
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 2.5 (5.5) | 7.0 (13.8) | 5.3 (6.5)

71. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 14
Description: as for outcome 68
Time Frame: as for outcome 5
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 3.8 (4.0) | 7.1 (10.3) | 6.7 (8.0)

72. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 16
Description: as for outcome 68
Time Frame: as for outcome 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
score on a scale | 2.5 (5.8) | 3.0 (6.2) | 6.0 (8.1)

73. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 20
Description: as for outcome 68
Time Frame: as for outcome 7
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | 1.9 (6.5) | 3.4 (10.7) | 3.6 (6.9)

74. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 24
Description: as for outcome 68
Time Frame: as for outcome 8
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | 2.1 (5.9) | 1.6 (5.7) | 6.1 (7.4)

75. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 28
Description: as for outcome 68
Time Frame: as for outcome 9
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
score on a scale | 4.3 (5.8) | 1.1 (8.0) | 3.6 (7.4)

76. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 32
Description: as for outcome 68
Time Frame: as for outcome 10
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 6
score on a scale | 2.9 (5.7) | 1.8 (6.1) | 7.7 (9.5)

77. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Week 34
Description: as for outcome 68
Time Frame: as for outcome 1
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 5
score on a scale | 5.6 (6.7) | 0.0 (8.6) | 6.4 (10.9)

78. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 12
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 6 | 5
score on a scale | 3.5 (7.1) | 0.7 (7.9) | 6.4 (10.9)

79. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 8
Description: The IBDQ Social Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | 1.3 (3.6) | 0.0 (2.4) | 0.7 (3.7)

80. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 10
Description: as for outcome 79
Time Frame: as for outcome 3
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | 2.5 (3.0) | 2.1 (4.7) | 1.1 (3.4)

81. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 12
Description: as for outcome 79
Time Frame: as for outcome 4
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | 3.0 (3.1) | 2.6 (5.1) | 2.3 (4.0)

82. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 14
Description: as for outcome 79
Time Frame: as for outcome 5
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | 2.8 (2.6) | 2.7 (3.4) | 4.0 (2.0)

83. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 16
Description: as for outcome 79
Time Frame: as for outcome 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
score on a scale | 2.5 (2.1) | 0.0 (3.9) | 2.4 (2.1)

84. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 20
Description: as for outcome 79
Time Frame: as for outcome 7
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 10 | 7 | 7
score on a scale | 2.8 (2.3) | 1.6 (3.0) | 3.6 (2.3)

85. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 24
Description: as for outcome 79
Time Frame: as for outcome 8
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 7 | 7
score on a scale | 1.8 (2.7) | -0.9 (4.9) | 2.6 (2.1)

86. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 28
Description: as for outcome 79
Time Frame: as for outcome 9
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 7 | 7
score on a scale | 2.1 (2.7) | -1.0 (4.6) | 2.4 (3.1)

87. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 32
Description: as for outcome 79
Time Frame: as for outcome 10
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 5 | 6
score on a scale | 1.3 (3.4) | -0.6 (2.9) | 3.3 (2.4)

88. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Week 34
Description: as for outcome 79
Time Frame: as for outcome 1
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 5 | 5
score on a scale | 3.0 (3.0) | 0.0 (3.4) | 3.0 (3.1)

89. Secondary Outcome: Change From Week 0 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 12
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 10 | 6 | 5
score on a scale | 1.7 (3.4) | -1.3 (4.5) | 3.0 (3.1)

90. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 0
Time Frame: Week 0 (relative to the start of the 6-week double-blind main study (N00291668)). 'Week 0' is the Baseline visit in the double-blind main study.
Population: Please see under the primary endpoint for explanation of entry into this extension study, C87048 (NCT00329420). Subjects who respond to re-induction in the Full Analysis Set with data at this time-point are included. Data collected after receipt of rescue therapy in a study have been set to missing in that study.
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
mg/L | 19.58 [4.0 to 60.0] | 14.97 [10.0 to 25.0] | 26.45 [16.0 to 50.0]

91. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 8
Time Frame: as for outcome 23
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
mg/L | 22.06 [8.0 to 76.0] | 11.91 [4.0 to 41.0] | 16.70 [1.0 to 55.0]

92. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 10
Time Frame: as for outcome 24
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
mg/L | 7.76 [2.0 to 40.0] | 5.62 [3.0 to 13.0] | 12.01 [1.0 to 34.0]

93. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 12
Time Frame: as for outcome 25
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
mg/L | 7.82 [2.0 to 31.0] | 7.06 [3.0 to 14.0] | 13.39 [1.0 to 54.0]

94. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 14
Time Frame: as for outcome 26
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
mg/L | 9.57 [2.0 to 32.0] | 6.32 [4.0 to 14.0] | 15.30 [1.0 to 41.0]

95. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 16
Time Frame: as for outcome 27
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
mg/L | 12.54 [3.0 to 35.0] | 12.23 [3.0 to 45.0] | 15.10 [1.0 to 36.0]

96. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 20
Time Frame: as for outcome 28
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
mg/L | 12.27 [1.0 to 74.0] | 13.24 [4.0 to 50.0] | 14.99 [1.0 to 53.0]

97. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 24
Time Frame: as for outcome 29
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
mg/L | 9.11 [1.0 to 45.0] | 14.16 [4.0 to 33.0] | 15.70 [1.0 to 38.0]

98. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 28
Time Frame: as for outcome 30
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
mg/L | 8.79 [1.0 to 24.0] | 14.25 [4.0 to 40.0] | 26.81 [0.0 to 33.0]

99. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 32
Time Frame: as for outcome 31
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 6
mg/L | 15.28 [3.0 to 45.0] | 10.27 [2.0 to 24.0] | 16.71 [1.0 to 48.0]

100. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 34
Time Frame: as for outcome 32
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 5
mg/L | 9.19 [1.0 to 40.0] | 6.23 [2.0 to 16.0] | 23.52 [0.0 to 81.0]

101. Secondary Outcome: C-Reactive Protein (CRP) Level at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Time Frame: as for outcome 33
Population: as for outcome 90
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 6 | 5
mg/L | 11.25 [1.0 to 75.0] | 8.46 [2.0 to 39.0] | 23.52 [0.0 to 81.0]

102. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 8 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 8 divided by the CRP Level at Week 0
Time Frame: as for outcome 2
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
ratio | 1.13 [0.4 to 4.3] | 0.80 [0.2 to 4.1] | 0.63 [0.0 to 3.4]

103. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 10 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 10 divided by the CRP Level at Week 0
Time Frame: as for outcome 3
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
ratio | 0.4 [0.1 to 1.5] | 0.38 [0.1 to 1.2] | 0.45 [0.0 to 2.0]

104. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 12 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 12 divided by the CRP Level at Week 0
Time Frame: as for outcome 4
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
ratio | 0.4 [0.1 to 2.0] | 0.47 [0.2 to 1.1] | 0.51 [0.0 to 3.2]

105. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 14 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 14 divided by the CRP Level at Week 0
Time Frame: as for outcome 5
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
ratio | 0.49 [0.1 to 5.0] | 0.42 [0.2 to 1.0] | 0.58 [0.0 to 2.4]

106. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 16 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 16 divided by the CRP Level at Week 0
Time Frame: as for outcome 6
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
ratio | 0.64 [0.1 to 5.3] | 0.82 [0.3 to 4.1] | 0.57 [0.0 to 2.3]

107. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 20 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 20 divided by the CRP Level at Week 0
Time Frame: as for outcome 7
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 7 | 7
ratio | 0.64 [0.0 to 5.5] | 0.88 [0.3 to 4.5] | 0.57 [0.0 to 3.1]

108. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 24 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 24 divided by the CRP Level at Week 0
Time Frame: as for outcome 8
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
ratio | 0.48 [0.0 to 3.5] | 0.95 [0.4 to 2.4] | 0.59 [0.0 to 1.7]

109. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 28 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 28 divided by the CRP Level at Week 0
Time Frame: as for outcome 9
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 7 | 7
ratio | 0.46 [0.0 to 2.8] | 0.95 [0.2 to 2.7] | 1.06 [0.0 to 2.1]

110. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 32 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 32 divided by the CRP Level at Week 0
Time Frame: as for outcome 10
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 6
ratio | 0.90 [0.1 to 4.6] | 0.64 [0.2 to 1.2] | 0.62 [0.0 to 2.8]

111. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 34 to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Week 34 divided by the CRP Level at Week 0
Time Frame: as for outcome 1
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 5 | 5
ratio | 0.54 [0.0 to 2.8] | 0.39 [0.2 to 1.6] | 1.07 [0.0 to 3.5]

112. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals) to CRP Level at Week 0
Description: The ratio is calculated as the C-Reactive Protein (CRP) Level at Last Visit (Week 34 for completers or the Withdrawal Visit for premature withdrawals)divided by the CRP Level at Week 0
Time Frame: as for outcome 12
Population: as for outcome 35
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 11 | 6 | 5
ratio | 0.59 [0.0 to 2.8] | 0.54 [0.2 to 2.8] | 1.07 [0.0 to 3.5]

113. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 8
Description: 70-point responders are subjects achieving a reduction in Crohn's Disease Activity Index (CDAI) score of ≥70 points from Week 0. CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
Time Frame: as for outcome 2
Population: Please see under the primary endpoint for explanation of entry into this extension study, C87048 (NCT00329420), and of 26 subjects being in the subgroup of "Responders to Re-induction", based on the Full Analysis Set. This explanation also details withdrawal or rescue therapy being counted as non-response from that time onwards in that study.
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 33.3 | 28.6 | 42.9
  Percentage of 70-point non-responders | 66.7 | 71.4 | 57.1

114. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 10
Description: as for outcome 113
Time Frame: as for outcome 3
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 66.7 | 85.7 | 100.0
  Percentage of 70-point non-responders | 33.3 | 14.3 | 0.0

115. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 12
Description: as for outcome 113
Time Frame: as for outcome 4
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 75.0 | 71.4 | 85.7
  Percentage of 70-point non-responders | 25.0 | 28.6 | 14.3

116. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 14
Description: as for outcome 113
Time Frame: as for outcome 5
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 100.0 | 100.0 | 100.0
  Percentage of 70-point non-responders | 0.0 | 0.0 | 0.0

117. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 16
Description: as for outcome 113
Time Frame: as for outcome 6
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 83.3 | 57.1 | 100.0
  Percentage of 70-point non-responders | 16.7 | 42.9 | 0.0

118. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 20
Description: as for outcome 113
Time Frame: as for outcome 7
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 75.0 | 71.4 | 85.7
  Percentage of 70-point non-responders | 25.0 | 28.6 | 14.3

119. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 24
Description: as for outcome 113
Time Frame: as for outcome 8
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 50.0 | 71.4 | 100.0
  Percentage of 70-point non-responders | 50.0 | 28.6 | 0.0

120. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 28
Description: as for outcome 113
Time Frame: as for outcome 9
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 58.3 | 71.4 | 85.7
  Percentage of 70-point non-responders | 41.7 | 28.6 | 14.3

121. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 32
Description: as for outcome 113
Time Frame: as for outcome 10
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 41.7 | 57.1 | 57.1
  Percentage of 70-point non-responders | 58.3 | 42.9 | 42.9

122. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Week 34
Description: as for outcome 113
Time Frame: as for outcome 1
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 66.7 | 42.9 | 42.9
  Percentage of 70-point non-responders | 33.3 | 57.1 | 57.1

123. Secondary Outcome: Percentage of Subjects Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0 at Last Visit (Week 34 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: as for outcome 113
Time Frame: as for outcome 12
Population: as for outcome 113
Measure: Number; unit: percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
percentage of subjects
  Percentage of 70-point responders | 66.7 | 42.9 | 42.9
  Percentage of 70-point non-responders | 33.3 | 57.1 | 57.1

124. Post Hoc Outcome: Number of Subjects With Disease Progression
Description: Disease progression is defined as:
  * an increase from Week 14 of ≥100 points in Crohn's Disease Activity Index (CDAI) score and CDAI>175 points for at least 2 consecutive visits,
  * use of rescue therapy, or,
  * subject withdrawal from the study.
Time Frame: as for outcome 34
Population: Non-responders at Week 6 of Study C87037 (NCT00291668) could enter this extension study C87048 (NCT00329420). As it was not possible to calculate the time to disease progression (outcome measure 34) due to the very small number of subjects meeting this definition, the post-hoc outcome of number of subjects with disease progression is presented here
Measure: Number; unit: subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 12 | 7 | 7
subjects | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data summarized in the first four columns were collected from the day after the end of the double-blind main study up to and including 12 weeks following the last dose received in this extension study for each subject (i.e., up to 36 weeks).
Description: For the fifth column, 'Total 2', this presents the data summarized in 'Total 1' PLUS adverse event data from the double-blind main study for subjects who received certolizumab pegol (CZP) in the main study and then entered this extension study (i.e., up to 44 weeks).
Groups:
- Total 1 (This Extension Study Only): This includes all adverse event data collected in this extension study for all 46 subjects who entered this extension study.
- Total 2 (Treatment With CZP in Main Study and Extension Study): This includes all adverse event data from the 6-week double-blind main study (N00291668) and this extension study for all 46 subjects who entered this extension study C87048, whilst they were receiving treatment with certolizumab pegol (CZP) in either study. Adverse events recorded in the double-blind main study (NCT00291668) for subjects who received Placebo treatment during that study are not included here.
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg | Total 1 (This Extension Study Only) | Total 2 (Treatment With CZP in Main Study and Extension Study)
Serious Adverse Events (participants affected / at risk) | 1/18 | 3/13 | 4/15 | 8/46 | 8/46
Other Adverse Events (participants affected / at risk) | 15/18 | 10/13 | 13/15 | 38/46 | 40/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CZP 400 mg / Placebo (N=18) | CZP 400 mg / CZP 200 mg (N=13) | CZP 400 mg / CZP 400 mg (N=15) | Total 1 (This Extension Study Only) (N=46) | Total 2 (Treatment With CZP in Main Study and Extension Study) (N=46)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 4 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Osteomalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Perianal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tetany (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CZP 400 mg / Placebo (N=18) | CZP 400 mg / CZP 200 mg (N=13) | CZP 400 mg / CZP 400 mg (N=15) | Total 1 (This Extension Study Only) (N=46) | Total 2 (Treatment With CZP in Main Study and Extension Study) (N=46)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
DNA antibody positive (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Dental caries (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Emotional distress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 2 (4)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site eyrthema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (2)
Nasopharyngitis (Infections and infestations) | 10 (15) | 5 (8) | 6 (7) | 21 (30) | 24 (39)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 5 (6)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Perianal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 6 (9) | 3 (3) | 11 (14) | 12 (16)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 5 (7)
White blood cell count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (2)

LIMITATIONS AND CAVEATS:
Due to the small number of subjects in this study, the percentages of subjects with adverse events may be misleading.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.